CLINICAL TRIAL: NCT07096596
Title: Understanding the Experiences and Challenges of People Living With Prostate Cancer
Brief Title: Prostate Cancer Study of Patient Experiences
Acronym: PROSPEX
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Yüksel Ürün, Professor doctor, Ankara University
Other Study IDs: ANKARA-UNIVERSITY-YURUN-001
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; survey; patient experience; oncology; health disparities; patient-reported outcomes; cancer care
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prostate Cancer Patients: Individuals diagnosed with prostate cancer, regardless of disease stage or treatment status. This group includes patients from diverse backgrounds and healthcare settings who are willing to share their experiences, challenges, and needs related to living with prostate cancer.
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No Intervention: Observational Cohort

SUMMARY:
The PROSPEX (PROstate cancer Study of Patient EXperiences) survey is designed to systematically assess the lived experiences, challenges, and unmet needs of individuals diagnosed with prostate cancer. This observational study will collect patient-reported data on psychological, social, and practical aspects of living with prostate cancer, including the impact on quality of life and access to care. The findings aim to inform the development of patient-centered interventions and improve supportive care strategies in future clinical trials and routine practice.

DETAILED DESCRIPTION:
Prostate cancer is one of the most common cancers among men worldwide, and its impact extends far beyond medical treatment, affecting many aspects of patients' lives. The PROSPEX (PROstate cancer Study of Patient EXperiences) project is designed to systematically capture the real-world experiences, challenges, and needs of individuals living with prostate cancer across diverse healthcare settings and backgrounds.

Objectives

The primary objectives of the PROSPEX study are:

1. To gather comprehensive, patient-reported data on the psychological, social, and practical challenges faced by people with prostate cancer, including the impact on quality of life, relationships, work, and daily living.
2. To identify disparities in access to care, supportive services, and information, as well as differences in patient experiences based on disease stage, treatment history, and demographic factors.
3. To inform the development of patient-centered care strategies and support services by highlighting unmet needs and areas for improvement in prostate cancer care.

Methods

The PROSPEX survey is an international, anonymous, online questionnaire designed for patients who have been diagnosed with prostate cancer. The survey includes between 70 and 125 questions, depending on each participant's disease stage and treatment history. It covers a wide range of topics, including demographic and clinical information, emotional well-being, social support, financial concerns, experiences with the healthcare system, and the impact of prostate cancer on daily life. The survey is expected to take approximately 30 to 60 minutes to complete. Participation is entirely voluntary, and no sensitive personal data or contact information will be collected or used. The study is investigator-initiated and receives no external funding; the research team declares no conflicts of interest.

Data Analysis Plan

Survey responses will be analyzed using both descriptive and inferential statistical methods. Comparative analyses will be conducted to identify variations in patient experiences across different regions, healthcare systems, and demographic groups. Advanced statistical techniques, such as regression analysis, may be used to explore factors associated with differences in quality of life, access to care, and patient outcomes.

Expected Impact

By systematically documenting the lived experiences of prostate cancer patients worldwide, the PROSPEX project aims to provide valuable insights into the challenges and unmet needs faced by this population. The findings are expected to inform healthcare providers, policymakers, and advocacy groups, guiding the development of more effective, patient-centered care and support services. Ultimately, PROSPEX seeks to improve the quality of life and care outcomes for individuals living with prostate cancer and to contribute to the global understanding of patient experiences in this disease.

ELIGIBILITY:
Inclusion Criteria:

Adults (aged 18 years or older). Diagnosed with prostate cancer at any stage (localized, locally advanced, metastatic, or recurrent).

Able to understand and provide informed consent for participation. Willing and able to complete the online survey in the available languages. Access to the internet and a device to complete the survey.

Exclusion Criteria:

Individuals who have not been diagnosed with prostate cancer. Individuals under 18 years of age. Inability to provide informed consent. Inability to complete the survey due to cognitive, language, or technical barriers.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult individuals (aged 18 and above) who have been diagnosed with prostate cancer, regardless of disease stage or treatment status. Participants will be recruited internationally and will represent a diverse range of backgrounds, healthcare settings, and geographic regions. The study aims to include patients with varying experiences, including those currently undergoing treatment, those in remission, and those living with advanced or recurrent disease. All participants must be able to provide informed consent and complete the online survey.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Characterization of global disparities in patient-reported experiences and quality of life among individuals with prostate cancer | One month
  Comparative analyses will be performed using survey data to identify and quantify differences in patient experiences, quality of life, and unmet needs across various regions and healthcare settings. Results will be reported as percentages of respondents, with thorough evaluation of territorial, institutional, and socioeconomic differences. Participants will be categorized according to the World Bank's income classification: low- and lower-middle-income countries, upper-middle-income countries, and high-income countries. Descriptive statistics will be used to compare demographic and clinical characteristics, as well as patient-reported outcomes. For categorical data, Pearson Chi-Square or Fisher's Exact test will be applied; for continuous variables, ANOVA will be used. A p-value of less than 0.05 will be considered statistically significant.

SECONDARY OUTCOMES:
Identification of factors associated with reduced quality of life and increased psychosocial burden in prostate cancer patients | one month
  Multivariate analyses, including regression modeling, will be conducted to explore associations between demographic, clinical, and healthcare system variables and patient-reported outcomes such as emotional well-being, social support, and financial concerns.
Assessment of disparities in access to supportive care and information among prostate cancer patients | one month
  Survey responses will be analyzed to determine differences in access to supportive services, information resources, and patient education across different regions and healthcare systems.

CONTACTS AND LOCATIONS:
Overall Officials: Yüksel Ürün, Study Director — Ankara University
Locations (1):
- Ankara University Faculty of Medicine, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the study director upon reasonable request.